CLINICAL TRIAL: NCT02987244
Title: Chidamide Plus CHOEP Combined With Upfront ASCT in Untreated Peripheral T-cell Lymphoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Chinese PLA General Hospital (Other); Peking University First Hospital (Other); Peking University Third Hospital (Other); Peking University Cancer Hospital & Institute (Other); Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-NHL-002
Record Dates: First submitted 2016-12-02; First posted 2016-12-08 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: T Cell Non-Hodgkin's Lymphoma
Keywords: Chidamide, T Cell Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Cyclophosphamide; Epirubicin; Vindesine; Etoposide; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- C-CHOEP (Experimental): experimental arm will be treated by Chidamide combined CHOEP ( cyclophosphamide, epirubicine, vindesine, etoposide and prednisone) regimen for 6 cycles.
  Interventions: Drug: Chidamide; Drug: Cyclophosphamide; Drug: Epirubicin; Drug: Vindesine; Drug: Etoposide; Drug: Prednisone

INTERVENTIONS:
Drug: Chidamide — Six cycles of therapy will be administered,and each cycle of treatment is 28 days.
  Phase I: Patients were treated at the following dose levels: 15, 20, and 25 mg twice per week to determine the MDT Phase II: If MTD was not reached at 25mg dose level of Chidamide. The followed study will use 20mg twice per week as experimental dose.
  Other Names: epidaza
Drug: Cyclophosphamide — Cyclophosphamide(750mg/m2) was administered intravenously on d1
Drug: Epirubicin — epirubicin (70mg/m2)was administered intravenously on d1;
Drug: Vindesine — vindesine (4mg)was administered intravenously on d1;
Drug: Etoposide — etoposide (100mg) was administered intravenously on d1,2,3.
Drug: Prednisone — prednisone (60mg/m2)was administered intravenously by oral d1-5.

SUMMARY:
The purpose of this study is to determine determine the maximum tolerated dose (MTD) and safety of the combination of Chidamide combined with CHOEP(cyclophosphamide， epirubicin,vindesine, etoposide and prednisone) regimen as first line treatment in newly-diagnosed T-NHL.

DETAILED DESCRIPTION:
Chidamide+Cyclophosphamide+Epirubicin+Vindesine+Etoposide+Prednisone Six cycles of therapy administered every 28 days were planned. Cyclophosphamide 750mg/m2 IV d1; epirubicin 70mg/m2 IV d1; Vindesine 4mg IV d1; etoposide 100mg IV d1-3; prednisone 60mg/m2 PO d1-5.

Chidamide:

Phase I: Patients were treated at the following bortezomib dose levels: 15, 20, and 25 mg twice per week.

Dose escalation and reduction were on the basis of the continual reassessment method, with at least two patients per dose level and no dose level skipped. No intrapatient dose escalation will be allowed. If one patient experienced dose-limiting toxicity (DLT), three additional patients were added to the dose level. If two of six patients experienced DLT, the previous dose level was declared the MTD. If only one of six patients experienced DLT, dose escalation was permitted to continue. DLT refers only to toxic events that occur during the first cycle of treatment.

At least 9(3+3+3) patients will be enrolled in Phase I study. Phase II: If MTD was not reached at 25mg dose level of Chidamide. The followed study will use 20mg twice per week as experimental dose.

After 3 Cycles, patients who become PD should withdraw the trial and receive other regimens; patients who become CR and eligible for auto-SCT will undergo auto-SCT; patients who get PR will receive 3 more cycles C-CHOEP regimen treatment, CR patients in them undergo auto-SCT, non-CR patients undergo follow-up phase.

All the patients will continue to receive chidamide treatment until progression of the disease (PD), unacceptable toxicity, or patient/investigator discretion.

During follow-uo phase, surveillance imaging with CT scans can be performed every 6 months up to the first 2 years, followed by doctor visit every 6 months up to 5 years or the disease relapses.

from recruiting the first subject until the last recruited subject finished his 2 years follow-up phase or the disease relapsed

ELIGIBILITY:
Inclusion Criteria:

* Newly-diagnosed T cell non-Hodgkin's lymphoma patients. Diagnosis of T cell NHL was performed by morphologic analysis of tissue pathological specimens along with Immunohistochemistry (IHC)
* ECOG≤2
* At least one or more unidimensionally measurable lesions (≥1 cm by CT scan or skin lesions or a measurable lesion by physical examination)
* Sign the Informed consent
* Women of childbearing potential must understand that the study medication could have a potential teratogenic risk. They should undergo complete contraception during the study period.
* Male subjects must agree to use condoms throughout study drug therapy.

Exclusion Criteria:

* T lymphoblastic leukemia/lymphoma
* Bone marrow involvement and lymphoma cell ≥ 25%
* Aplastic large T cell lymphoma - ALK positive
* NK/T-cell lymphoma
* Mycosis Fungoides/Sezary Syndrome
* Pre-existing uncontrolled active infection
* Clinical evidence of grade 3 or 4 heart failure as defined by the New York Heart Association criteria
* Grade 3 or 4 peripheral neuropathy
* Pregnancy or active lactation
* Co-existing tumors
* Impaired renal/ hepatic function (serum creatinine >1.5 mg/dl or creatinine clearance <60 ml/min or serum transaminases/ bilirubin ≥3 upper limits of normal）
* History of mental illness

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-03; Primary Completion 2020-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
2 years progression-free survival | the overall time frame is up to 48 months
  from recruiting the first subject until the last recruited subject finished his 2 years follow-up phase or the disease relapsed

SECONDARY OUTCOMES:
5 years overall survival（OS） | the overall time frame is up to 84 months
  from recruiting the first subject until the last recruited subject finished his 5 years follow-up phase
overall response rate(ORR) and complete remission rate(CR） | the overall time frame is up to 30 months
  the last recruited subject finished 4 cycle C-CHOEP regimen
adverse events | the overall time frame is up to 84 months
  throughout the treatment and until 30 days after the administration of the last dose of a study drug

OTHER OUTCOMES:
maximum tolerated dose of chidamide | the overall time frame is up to 6 months
  from recruiting the first 9 subjects to all of them received 1 cycle C-CHOEP regiment

CONTACTS AND LOCATIONS:
Overall Officials: Daobin Zhou, M.D, Principal Investigator — Peking Union Medical College Hospital
Locations (2):
- China (2):
  - Peking Union medical college hospital, Beijing, Beijing Municipality
  - Tianjin medical universty cancer institute & hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dong M, Ning ZQ, Xing PY, Xu JL, Cao HX, Dou GF, Meng ZY, Shi YK, Lu XP, Feng FY. Phase I study of chidamide (CS055/HBI-8000), a new histone deacetylase inhibitor, in patients with advanced solid tumors and lymphomas. Cancer Chemother Pharmacol. 2012 Jun;69(6):1413-22. doi: 10.1007/s00280-012-1847-5. Epub 2012 Feb 24. PMID 22362161
- [Background] Shi Y, Dong M, Hong X, Zhang W, Feng J, Zhu J, Yu L, Ke X, Huang H, Shen Z, Fan Y, Li W, Zhao X, Qi J, Huang H, Zhou D, Ning Z, Lu X. Results from a multicenter, open-label, pivotal phase II study of chidamide in relapsed or refractory peripheral T-cell lymphoma. Ann Oncol. 2015 Aug;26(8):1766-71. doi: 10.1093/annonc/mdv237. Epub 2015 Jun 23. PMID 26105599
- [Derived] Wang W, Zhang W, Su LP, Liu LH, Gao YH, Wang QS, Su H, Song YQ, Zhang HL, Shen J, Jing HM, Wang SY, Cen XN, Liu H, Liu AC, Li ZJ, Luo JM, He JX, Wang JW, O'Connor OA, Zhou DB. Efficacy of chidamide maintenance therapy versus autologous stem cell transplantation versus observation as a post-remission choice in the survival of adult patients with peripheral T-cell lymphoma: Post hoc analysis of a prospective, multicenter, phase 2 study in China. Ann Hematol. 2024 Aug;103(8):3061-3069. doi: 10.1007/s00277-024-05708-w. Epub 2024 May 28. PMID 38805037
- [Derived] Zhang Y, Zhang W, Li J, Duan M, Han B, Zhu T, Zhuang J, Cai H, Cao X, Chen M, Zhou D. Gemcitabine, cisplatin, and dexamethasone (GDP) in combination with methotrexate and pegaspargase is active in newly diagnosed peripheral T cell lymphoma patients: a phase 2, single-center, open-label study in China. Ann Hematol. 2019 Jan;98(1):143-150. doi: 10.1007/s00277-018-3488-1. Epub 2018 Sep 12. PMID 30209556